CLINICAL TRIAL: NCT01443507
Title: Does Endurance Exercise With Low Intensity and Longer Duration Improve Aerobic Capacity to the Same Extent as High Intensity Interval Training?
Brief Title: Effect of Exercise With Low Intensity and Longer Duration Versus High Intensity Interval Training
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Volda University College (Other)
Collaborators: helse Møre og Romsdal, Volda sjukehus (Unknown)
Responsible Party: Principal Investigator, Kjetil Laurits Hoydal, Phd, associate professor, Volda University College
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2010/2959
Record Dates: First submitted 2011-09-21; First posted 2011-09-29 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Subjects
Keywords: aerobic capacity; maximal oxygen uptake; aerobic endurance; work economy; lactate threshold; endurance training; exercise intensity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high intensity long interval (Experimental): A group training four by four minutes interval at 90-95% of maximal heart rate dispersed by three minutes active pauses at 70% of maximal heart rate.
  Interventions: Other: endurance exercise of different duration and intensity
- long duration at moderate training (Experimental): a continuous training group exercising at 70% of maximal heart rate for 90 minutes.
  Interventions: Other: endurance exercise of different duration and intensity

INTERVENTIONS:
Other: endurance exercise of different duration and intensity — Two interventions are compared with aerobic capacity as the main outcome. one group exercise at 70% of maximal heart rate for 90 minutes 3 times per week. group two exercise performe10 minutes warm up at 70% of maximal heart rate 4 x 4 minutes intervals at 90-95% of maximal heart rate with 3 minutes active pause at 70% of maximal heart rate in between, and finally 5 minutes cooling down at 70 % of maximal heart rate.

SUMMARY:
The purpose of the study is to compare exercise at 70% of maximal heart rate were total energy expenditure is twice compared to interval training at 90- 95% of maximal heart rate. Since 70% of maximal heart rate is well above the minimum threshold for improvements in maximal oxygen uptake it should be suited to investigate the effect of duration.

ELIGIBILITY:
Inclusion Criteria:

* healthy non smoking men and woman, age 18-30

Exclusion Criteria:

* pathological findings measured by ekko/doppler, high cholesterol or high blood pressure

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
changes in maximal oxygen uptake | Maximal oxygen uptake will be measured at day 1 before training, then we will measure changes in maximal oxygen uptake after 8 weeks, and finally a follow up measurement of changes in maximal oxygen uptake after 1 year

SECONDARY OUTCOMES:
endurance performance | one year
  work economy, lactate threshold will be measured toghether with maximal oxygen uptake to determine endurance performance.
health effects | one year
  coronary flow reserve, blood pressure, maximal oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Aud Folkestad, dean, Study Director — Volda University College
Locations (1):
- Volda university college, Volda, Volda, Norway